CLINICAL TRIAL: NCT05310331
Title: Efficacy and Safety of Donafenib Combined With Paclitaxel and Platinum in Patients With Recurrent, Metastatic, and Persistent Advanced Cervical Cancer: A Single-arm, Phase II Study
Brief Title: Donafenib for Recurrent Cervical Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DONA1
Record Dates: First submitted 2022-03-26; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Targeted Therapy; Chemotherapy; Recurrent Cervical Carcinoma; Metastatic Cervical Carcinoma; Persistent Advanced Cervical Carcinoma; Survival Outcomes; Adverse Effect
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with recurrent cervical cancer (Experimental): Eligible patients according to inclusion and exclusion criteria.
  Interventions: Combination Product: Donafenib combined with paclitaxel and platinum ± PD-1 antibody

INTERVENTIONS:
Combination Product: Donafenib combined with paclitaxel and platinum ± PD-1 antibody — Patients will receive Donafenib (200mg, bid) combined with paclitaxel (135mg/m2) and cisplatin (creatinine clearance rate > 60ml/min, 50 mg/m2) or paclitaxel (175 mg/m2) and carboplatin AUC=5 (40ml/min < creatinine clearance rate < 60ml/min) ± PD-1 antibody every 3 weeks.

SUMMARY:
This study is to evaluate the safety and tolerability of Donafenib combined with paclitaxel and platinum ± programmed death 1 monoclonal antibody (PD-1 antibody) in patients with recurrent cervical cancer.

DETAILED DESCRIPTION:
This is a single center, non-randomized, open-label Phase II clinical study to investigate the efficacy and tolerability of Donafenib combined with paclitaxel and platinum ± PD-1 antibody in patients with recurrent cervical cancer. In total 20 patients will receive Donafenib (200mg, bid) combined with paclitaxel (135mg/m2) and cisplatin (creatinine clearance rate > 60ml/min, 50 mg/m2) or paclitaxel (175 mg/m2) and carboplatin AUC=5 (40ml/min < creatinine clearance rate < 60ml/min) ± PD-1 antibody every 3 weeks.

Actual Study Start Date: March 27, 2022 Estimated Primary Completion Date: December 27, 2023 Estimated Study Completion Date: June 27, 2024

Arms There is only one arm, i.e., group of Donafenib combined with paclitaxel and platinum ± PD-1 antibody. Each treatment period was 21 days. Patients will be treated with 4-6 cycles of Donafenib plus TP or TC ± PD-1 antibody. After completion of the combination, patients will be maintained on Donafenib until disease progression or unacceptable toxicity occurs (up to 12 months)

Donafenib was taken orally at 200 mg twice on an empty stomach (1 hour before or > 2 hours after meal) in the morning and evening of each administration day, with an interval of about 12 hours. Maintain the same dose until disease progression, death, toxicity intolerance, withdrawal of informed consent, initiation of new antineoplastic therapy, or termination of treatment for other reasons specified in the protocol, for a maximum of 12 months.

Paclitaxel and platinum:

If creatinine clearance rate > 60ml/min: on Day 1 of each 21-day cycle, participants receive an intravenous (IV) infusion of paclitaxel 135 mg/m2plus cisplatin 50 mg/m2.

If 40ml/min < creatinine clearance rate < 60ml/min:on Day 1 of each 21-day cycle, participants receive an intravenous (IV) infusion of paclitaxel 175 mg/m2 plus carboplatin AUC=5.

PD-1 antibody: PD-1 antibody is not mandatory, intravenous infusion on the first day of each cycle, every 3 weeks for a cycle until disease progression, death, toxicity intolerance, withdrawal of informed consent, initiation of new antitumor therapy, or termination of treatment for other reasons specified in the protocol, the longest treatment period is 12 months.

The primary outcome measure is progression-free survival. The secondary outcome measures include overall survival, objective response rate, etc.

ELIGIBILITY:
Inclusion criteria

* Written informed consent obtained.
* Age 18~75, female.
* Histologically confirmed cervical squamous cell carcinoma, adenosquamous carcinoma or adenocarcinoma.
* Patients with cervical cancer recurred for the first time, and did not receive any treatment after recurrence.
* Patients must have measurable disease per RECIST 1.1.
* ECOG performance status 0 or 1, expected lifetime ≥ 3 months.
* No targeted drugs containing VEGF were used before, including but not limited to anlotinib, apatinib, bevacizumab, etc.
* Adequate organ function:
* Absolute neutrophil count (ANC) ≥ 1.5x109/L, Platelets ≥ 100x109/L, Hemoglobin (Hb) ≥ 90g/L, Bilirubin ≤ 1.5 times the upper limit of normal, ALT/AST ≤ 3x ULN (for patient with liver metastasis ALT/AST ≤ 5x ULN), Serum bilirubin ≤1.5x ULN, Serum creatinine ≤ 1.5 times the upper limit of normal, and creatinine clearance ≥ 40ml/min (calculated by Cockcroft-Gault formula); International normalized ratio (INR) ≤1.5

Exclusion Criteria:

* Histopathologic diagnoses of tumors other than squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma.
* With second primary malignant diseases.
* Pregnancy or children bearing potential.
* With uncontrolled auto-immune diseases, interstitial pneumonia, ulcerative colitis, or patients who should receive long-term glucocorticoid treatment (>10mg/d prednisone).
* With uncontrollable complications.
* Conditions which impact on pill taking (dysphagia, chronic diarrhea, bowel obstruction).
* Known hypersensitivity reaction to any of the study drugs or components.
* Other unsuitable conditions determined by investigators.
* Hepatitis B virus (HBV) >2000 IU/ml or DNA ≥ 1×10^4/ml; or hepatitis C virus (HCV) RNA ≥ 1×10^3/ml).
* Has received a live vaccine within 4 weeks prior to the first dose of trial treatment. Note: Injection of inactivated viral vaccines against seasonal influenza are allowed.
* Has pleural effusion and ascites that require punctured and drained. However, an exception includes patients with pleural effusion and ascites who have no symptoms.
* Any other medical, psychiatric, or social condition deemed by the investigator to be likely to interfere with a subject's rights, safety, welfare, or ability to sign informed consent, cooperate, and participate in the study or would interfere with the interpretation of the results.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-12-27 (Estimated); Study Completion 2024-06-27 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 24 months
  PFS defined as the time the duration from date of enrollment to the first documented disease progression, or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival | 36 months
  Overall survival is defined as the duration from date of enrollment to the date of death from any cause.
Objective Response Rate (ORR) | 24 months
  ORR is defined as the percentage of participants in the analysis population who have a complete or partial remission.
Duration of Response (DCR) | 24 months
  DCR is defined as the percentage of participants in the analysis population who have a complete or partial remission, or stable disease (SD).
Adverse Events | 24 months
  Adverse event (AE)、Treatment emergent adverse event (TEAE)、Serious adverse event (SAE).

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China